CLINICAL TRIAL: NCT05837403
Title: The Use of Platelet-rich Plasma in the Treatment of Chronic Anal Fissure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Al-Kindy College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14 Al-KindyCM
Record Dates: First submitted 2022-11-14; First posted 2023-05-01 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Fissure in Ano
Keywords: Fissure in Ano; Platelet-Rich Plasma; Lateral Internal Sphincterotomy
MeSH Terms: conditions — Fissure in Ano

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitroglycerin only (Active Comparator): application of local Nitroglycerin ointment 2% (Recto-Relief Nitroglycerin Ointment, 30 g) applied twice daily.
  Interventions: Drug: Nitroglycerin ointment
- platelet rich plasma injection (Experimental): injection of platelet rich plasma under fissure base and edges
  Interventions: Procedure: Platelet rich plasma injection; Drug: Nitroglycerin ointment

INTERVENTIONS:
Procedure: Platelet rich plasma injection — venous blood drown from the patient, centrifugation and separation of platelet rich plasma, injection under fissure and edges base.
  Arms: platelet rich plasma injection
Drug: Nitroglycerin ointment — application of the ointment twice daily
  Other Names: Rectocare - Ointment

SUMMARY:
use of platelet rich plasma had good effect in treating chronic wounds. healing of perianal fissure could be prolonged and associated with pain. injection of platelet rich plasma under fissure base and edges had the advantage of improved fissure healing and reduction of the pain, with minimal side effects.

DETAILED DESCRIPTION:
Thirty milliliters of venous blood were withdrawn into eight syringes with preloaded 0.4 milliliters of anticoagulant (dextrose solution A) in each syringe to achieve concentration of 9:1.

The mixture centrifuged for 3000 round per minute for three minutes. After centrifugation separation of supernatant from the red blood cells, using three way-stopcock connector to collect the supernatant of all syringes into four new syringes that preloaded with 1 microgram of Prostaglandin E1 that diluted in normal saline (0.05 milliliters).

The four syringes centrifuge at 4000 round per minute for 15 minutes. The supernatant discarded using a three way-stopcock connector. The sediment mixed with vortex mixer (Vortex V-1 plus, BIOSAN).

ELIGIBILITY:
Inclusion Criteria:

• chronic anal fissure for more than three months

Exclusion Criteria:

* medical comorbidity
* inflammatory bowel disease
* tuberculosis fissure
* HIV infected patients

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 460 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Healing of fissure | 3 months
  Complete epithelization of fissure base

SECONDARY OUTCOMES:
Duration of pain | 3 months
  Duration of pain after passing bowel motion measured in minutes
Pain change | 3 months
  Visual analog scale for measuring the intensity of pain (the higher score means the more severe the pain) explained as 0 represent no pain at all, and 10 represent the severest pain ever felt.

CONTACTS AND LOCATIONS:
Overall Officials: Taghreed Alhaidari, C.A.B.O.G, Study Chair — Al-Kindy College of Medicine
Locations (1):
- Al-Kindy Teaching Hospital, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No